CLINICAL TRIAL: NCT04498169
Title: A Randomized, Open-Label, Parallel-Group Study to Evaluate the Safety and Efficacy of Two Dosing Regimens of Netarsudil Ophthalmic Solution in Patients With Corneal Edema Due to Fuchs Corneal Dystrophy
Brief Title: A Phase 2 Study Evaluating the Safety and Efficacy of Netarsudil Ophthalmic Solution in Patients With Corneal Edema Due to Fuchs Corneal Dystrophy
Acronym: Fuchs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AR-13324-CS210
Record Dates: First submitted 2020-07-31; First posted 2020-08-04 (Actual); Results first posted 2022-09-01 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Corneal Edema
Keywords: Corneal Edema; Fuchs Corneal Dystrophy; Netarsudil Ophthalmic Solution
MeSH Terms: conditions — Corneal Edema; Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Once Daily Netarsudil Ophthalmic Solution (Experimental): One drop of Netarsudil 0.02% ophthalmic solution in the study eye in the evening for an 8 week period in up to 20 subjects.
  Interventions: Drug: Netarsudil Ophthalmic
- Twice Daily Netarsudil Ophthalmic Solution (Experimental): One drop of Netarsudil 0.02% ophthalmic solution in the study eye in the morning and in the evening for an 8 week period in up to 20 subjects.
  Interventions: Drug: Netarsudil Ophthalmic

INTERVENTIONS:
Drug: Netarsudil Ophthalmic — Netarsudil Ophthalmic Solution 0.02% Topical Sterile Ophthalmic Solution
  Other Names: Rhopressa®
  Arms: Once Daily Netarsudil Ophthalmic Solution
Drug: Netarsudil Ophthalmic — Netarsudil Ophthalmic Solution 0.02% Topical Sterile Ophthalmic Solution
  Other Names: Rhopressa®
  Arms: Twice Daily Netarsudil Ophthalmic Solution

SUMMARY:
Two different dosing regimens (QD and BID) of netarsudil will be studied to evaluate their efficacy in reducing or resolving corneal edema in subjects with FCD.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older
2. Documented diagnosis of FCD
3. Evidence of central corneal edema, in at least one eye, at the Screening and Baseline Visit, in the eligible eye(s)
4. Reduced BCVA secondary to central corneal edema, at Screening and Baseline, in the eligible eye(s)

Exclusion Criteria:

1. FCD so advanced that, in the opinion of the Investigator, surgery would likely be required in the study eligible eye(s) within the study period
2. Clinically significant ocular disease (other than FCD) or trauma in the eligible eye(s) which could interfere with study interpretation
3. History of ocular surgery within 6 months of the Screening Visit, or any prior corneal refractive surgery in the eligible eye(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Senchyna, Ph.D., Study Director — Aerie Pharmaceuticals Inc.
Locations (12):
- United States (12):
  - Orange County Ophthalmology, Garden Grove, California
  - Harvard Eye Associates, Laguna Hills, California
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Advance Eye Associates, South Dartmouth, Massachusetts
  - Chu Vision Institute, Bloomington, Minnesota
  - Minnesota Eye Care, Minnetonka, Minnesota
  - Ophthalmology Associates, St Louis, Missouri
  - Vance Thompson Vision, West Fargo, North Dakota
  - Comprehensive Eye Care, Westerville, Ohio
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Houston Eye Associates, Houston, Texas
  - Virginia Eye Consultants, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lindstrom RL, Lewis AE, Holland EJ, Sheppard JD, Hovanesian JA, Senchyna M, Hollander DA. Phase 2, Randomized, Open-Label Parallel-Group Study of Two Dosing Regimens of Netarsudil for the Treatment of Corneal Edema Due to Fuchs Corneal Dystrophy. J Ocul Pharmacol Ther. 2022 Dec;38(10):657-663. doi: 10.1089/jop.2022.0069. Epub 2022 Nov 3. PMID 36327101

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at 12 clinic sites in the United States between September 2020 and June 2021.
Pre-assignment Details: All participants underwent a washout of their pre-study treatment for Fuchs Corneal Dystrophy for a period of 24 hours prior to the baseline visit.
Groups:
- Once Daily Netarsudil Ophthalmic Solution: One drop of study artificial tear in the study eye in the morning, and one drop of Netarsudil 0.02% ophthalmic solution in the study eye in the evening for an 8 week period in up to 20 subjects.
  Netarsudil Ophthalmic: Netarsudil Ophthalmic Solution 0.02% Topical Sterile Ophthalmic Solution
Period: Modified Intent-to-Treat Population
Arm/Group | Once Daily Netarsudil Ophthalmic Solution | Twice Daily Netarsudil Ophthalmic Solution
Started | 20 | 20
Completed | 19 | 19
Not Completed | 1 | 1
Period: Safety Population
Arm/Group | Once Daily Netarsudil Ophthalmic Solution | Twice Daily Netarsudil Ophthalmic Solution
Started | 20 | 20
Completed | 19 | 19
Not Completed | 1 | 1
Period: Per-Protocol Population
Arm/Group | Once Daily Netarsudil Ophthalmic Solution | Twice Daily Netarsudil Ophthalmic Solution
Started | 18 | 16
Completed | 18 | 15
Not Completed | 0 | 1
Period: Study Completion
Arm/Group | Once Daily Netarsudil Ophthalmic Solution | Twice Daily Netarsudil Ophthalmic Solution
Started | 20 | 20
Completed | 19 | 19
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: 40 participants were randomized; 20 each to the Netarsudil QD and the Netarsudil BID arms. 1 participant discontinued from each arm due to adverse events.
  40 participants were included in both the mITT population for the primary endpoint analysis and the safety population for safety analysis.
  6 participants were excluded from the per-protocol analysis due to protocol deviations (2 in the Netarsudil QD arm, 4 in the Netarsudil BID arm). There were no Covid-19 related protocol deviations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Once Daily Netarsudil Ophthalmic Solution | Twice Daily Netarsudil Ophthalmic Solution | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 11 | 11 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 11 | 8 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 0 | 2 | 2
  White | 20 | 18 | 38
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Central Corneal Thickness (CCT)
Description: Mean change from baseline in CCT by ultrasound pachymetry
Time Frame: Baseline & 4 weeks
Population: Modified Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Once Daily Netarsudil Ophthalmic Solution | Twice Daily Netarsudil Ophthalmic Solution
Number analyzed (Participants) | 20 | 20
µm | -28.4 (35.72) | -20.1 (39.12)
Statistical Analysis 1: Comparison: Once Daily Netarsudil Ophthalmic Solution vs Twice Daily Netarsudil Ophthalmic Solution; The primary analysis used the mITT population with available data per subject at eye level (ie., ODO). Robustness analyses was also performed based on the MI methodology under different assumptions of missingness and intercurrent events (where missing data or withdrawal due to lack of efficacy or AEs were imputed using FCS regression method and missing data for all other reasons were imputed using worst within subject observation prior to the intercurrent event); Test type: Superiority — With a sample size of up-to 20 subjects within a treatment group, the study had 80% power to demonstrate a statistically significant mean change from baseline, assuming the true effect size (mean change / SD) was 0.577 or larger (e.g. assuming the true mean change from baseline was 34.6 μm and the SD was 60 μm), a one sample t-test and a two-sided alpha = 0.10; p = 0.0021, One-sample t-test (within group)

ADVERSE EVENTS:
Time Frame: Adverse events were documented from the time of signing the informed consent until the last study visit for each participant. This was a period of approximately 8 weeks (56 days) for participants who completed the full study duration. For AEs ongoing at the time of study completion, the ongoing AE was followed-up and the participant was provided appropriate medical care until the event resolved or stabilized, the participant was lost to follow-up, or there was other resolution to the event.
Description: Adverse events information was collected at all study visits.
Arm/Group | Once Daily Netarsudil Ophthalmic Solution | Twice Daily Netarsudil Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 5/20 | 7/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Once Daily Netarsudil Ophthalmic Solution (N=20) | Twice Daily Netarsudil Ophthalmic Solution (N=20)
Viral gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Once Daily Netarsudil Ophthalmic Solution (N=20) | Twice Daily Netarsudil Ophthalmic Solution (N=20)
Corneal verticillata (Eye disorders) | 3 (3) | 2 (2)
Conjunctival hypaeremia (Eye disorders) | 2 (4) | 4 (4)
Erythema of eyelid (Eye disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT04498169/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT04498169/SAP_001.pdf